CLINICAL TRIAL: NCT03152565
Title: A Single Arm Phase I-II Multicenter Trial With Avelumab Plus Autologous Dendritic Cell Vaccine to Determine Safety and Preliminary Efficacy of the Combination in Pre-treated Mismatch Repair-proficient (MSS) Metastatic Colorectal Cancer Patients.
Brief Title: Avelumab Plus Autologous Dendritic Cell Vaccine in Pre-treated Metastatic Colorectal Cancer Patients
Acronym: AVEVAC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-1602; 2016-003838-24 (EudraCT Number)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab in combination ADC vaccine (Experimental): Patients in both phases will receive Avelumab biweekly intravenous during a maximum of 12 months and biweekly 10x106 ADC vaccine (intradermal) for five doses (days 1, 14, 28, 42 and 56) followed by a maximum of 6 doses every 6 months.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Autologous Dendritic Cells vaccine: A dose of ADC at days 1, 14, 28, 42 and 56 (total of 5 doses), and thereafter every 6 months until disease progression (maximum of 6 additional doses) or unacceptable toxicity.
  Avelumab will be administered intravenously at a dose of 10 mg per kilogram of body weight, every 14 days until disease progression or unacceptable toxicity.
  Other Names: Autologous Dendritic Cells

SUMMARY:
Single arm Phase I/II multicentric open labeled, with translational sub-study, of avelumab plus autologous dendritic cell vaccine in pre-treated mismatch repair-proficient (MSS) metastatic colorectal cancer patients..

DETAILED DESCRIPTION:
This 2-phases study will first evaluate two different doses/schema of avelumab plus autologous dendritic cell vaccine (ADC) vaccines, in intention to define which dose is effective without hampering safety. Second phase will consist in an standard analysis of efficacy and progression free survival. It is expected that 4 Spanish Sites will include patients in phase I and 8 Spanish Centers will include patients in the phase II of the study

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of approved by the investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to the performance of any trial activities.
* Histological diagnosis of MSS colorectal adenocarcinoma.
* Metastatic disease treated with at least two chemotherapy line, with or without targeted therapies.
* Male or female subjects aged ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.
* Lactate dehydrogenase (LDH) levels (<1.5 ULN) (between 250-450 U/L). Maximum allowed 675 U/L.
* Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normality (ULN) and Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
* Negative serum pregnancy test at screening for women of childbearing potential.
* Highly effective contraception for both male and female subjects throughout the study and for at least 60 days after last avelumab treatment administration if the risk of conception exists.
* Adequate hematological function: a) Haemoglobin ≥ 9 g/dL (may have been transfused).

  b) Platelet count ≥ 100 × 109/L. c) Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
* Renal: Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.

Exclusion Criteria:

* Subjects with brain metastases.
* Prior organ transplantation, including allogeneic stem-cell transplantation.
* Presence of clinical ascites.
* Modified Charlson score >2 (excluded cancer).
* Significant acute or chronic infections including, among others: Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Positive test for Hepatitis C Virus (HCV) surface antigen and / or confirmatory Hepatitis C Virus (HCV) Ribonucleic acid (RNA) (if anti-HCV antibody tested positive).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent: a)Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible. b) Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg/24 h of prednisone or equivalent. c) Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intraocular, or inhalation) are acceptable.
* Local positive serologic determination to: Hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (Anti-HBc), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), HCV ribonucleic acid test (HCV RNA), HIV-I RNA, Agp24 III-V + Carbonic anhydrase III-V (CAIII-V) ½ (MLIA) serum, Immunoglobulin G (Ig) antigen core HBV, reaginic antibodies (RPR) for Systemic Erythematosus Lupus (SEL-RPR) serum, immunoglobulin G (IgG), cytomegalovirus (EIA), Anti-Human T-Cell Lymphotropic I/II Viruses (HTLV) Antigens (if patient came from endemic zone), Anti-Trypanosoma Cruzi antibodies, Chagas (if patient came from endemic zone), when RPR positive or doubtful for confirmation: IgG Treponema pallidum (ELISA), Immunoglobulin M (IgM) Treponema pallidum (ELISA), when IgG T. Pallidum doubtful: Pt confirmatory IgG/IgM, Treponema pallidum (LIA).
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 according National Cancer Institute-Common Terminology for Common Adverse Events/NCI-CTCAE v 4.03), - any history of anaphylaxis, or uncontrolled asthma. Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy Grade ≤ 2 is acceptable.
* Pregnancy or lactation.
* Known alcohol or drug abuse.
* All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment
* Any psychiatric condition that would impede the understanding of informed consent
* Vaccination other study treatment is prohibited, within 4 weeks of the first dose of avelumab and while on trial.
* History of other tumors in the past 5 years.
* Active infections.
* Current immunosuppressive treatment, except for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)."
* Known hypersensitivity to avelumab, ADC vaccines or their components.
* Legal incapacity or limited legal capacity.
* Patients with pneumonitis and pulmonary fibrosis.
* Patients with cardiac medical history: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 180 days after the last dose of ADC + avelumab combination therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Dose of Avelumab in combination with Autologous Dendritic Cells | 18 months
  Dose of avelumab at which no dose limiting toxicity is shown.
Progression Free Survival | 6 months
  Percentage of patients without progression of disease

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 18 months
  Frequency, nature and number of patients developing adverse events throughout follow up
Modified Consensus Molecular Subtypes' (CMS) classification of Immunophenotype signature in tumor biopsies before and during treatment. | 18 months
  Modified CMS classification by NanoString
Immunophenotype signature in tumor biopsies before and during treatment. | 18 months
  MSS, RAS and BRAF mutation status at baseline and during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Maurel Santasusana, M.D., Principal Investigator — Hospital Clinic of Barcelona
Locations (8):
- Spain (8):
  - Hospital Clínic Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espanol-Rego M, Fernandez-Martos C, Elez E, Foguet C, Pedrosa L, Rodriguez N, Ruiz-Casado A, Pineda E, Cid J, Cabezon R, Oliveres H, Lozano M, Gines A, Garcia-Criado A, Ayuso JR, Pages M, Cuatrecasas M, Torres F, Thomson T, Cascante M, Benitez-Ribas D, Maurel J. A Phase I-II multicenter trial with Avelumab plus autologous dendritic cell vaccine in pre-treated mismatch repair-proficient (MSS) metastatic colorectal cancer patients; GEMCAD 1602 study. Cancer Immunol Immunother. 2023 Apr;72(4):827-840. doi: 10.1007/s00262-022-03283-5. Epub 2022 Sep 9. PMID 36083313